CLINICAL TRIAL: NCT06722482
Title: Clinical Evaluation of Freeze-Dried Bone Allograft Compared to Collagen-Enriched Bovine Xenograft for Alveolar Ridge Preservation of Anterior Extraction Sockets.
Brief Title: Comparison of Two Types of Bone Grafts in Patients Who Need One of Their Front Teeth Removed and Replaced With an Implant
Acronym: FDBA or CEBX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Implant Dentistry Research & Education Foundation (IDREF) (Unknown)
Responsible Party: Principal Investigator, Elli Kotsailidi, Assistant professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008216; AWD00006192 (Other Grant/Funding Number: Implant Dentistry Research & Education Foundation (IDREF))
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ridge Preservation; Allografts; Extraction, Tooth; Xenograft
Keywords: alveolar ridge preservation; tooth extraction; freeze-dried bone allograft; collagen-enriched bovine xenograft

STUDY DESIGN:
Intervention Model Description: single center, pilot, randomized, clinical trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded in regards to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FDBA arm (Experimental)
  Interventions: Device: FDBA
- CEBX arm (Active Comparator)
  Interventions: Device: CEBX

INTERVENTIONS:
Device: FDBA — Twenty five participants will receive FDBA in anterior extraction sockets as part of the alveolar ridge preservation procedure.
  Other Names: Freeze-dried bone allograft
  Arms: FDBA arm
Device: CEBX — Twenty five participants will receive CEBX in anterior extraction sockets as part of the alveolar ridge preservation procedure.
  Other Names: Collagen-enriched bovine xenograft
  Arms: CEBX arm

SUMMARY:
The purpose of this study is to compare two different bone graft materials (freeze-dried bone allograft, FDBA and collagen-enriched bovine xenograft, CEBX) that are routinely used for preserving the remaining bone after extraction of an anterior tooth, and before placing a dental implant. Patients will be randomly assigned to either group (flip of a coin) One group will receive FDBA material and the other group will receive CEBX (cow) material.

The study aims to examine the following main questions:

* Potential differences in linear radiographic horizontal (HRD) and vertical (VRD) ridge dimensional changes between groups after 16 weeks of healing
* Other clinical information of the treated areas and information regarding the esthetics of the dental implant that will subsequently be placed at the edentulous site as well as patient satisfaction with the treatment, will be evaluated.

The study will include 7 study visits. Study procedures will take place during the same visits as the standard of care treatments (tooth extraction and bone graft, dental implant placement, crown installation and follow-ups). Clinical information from these standard of care visits will be used for the current research study, such as:

* Demographic information
* Clinical information from intraoral photographs
* Radiographic information from cone beam computed tomography and periapical radiographs.

DETAILED DESCRIPTION:
The study will compare clinical, radiographic (dental cone beam computed tomography) and histologic outcomes upon tooth extraction and alveolar ridge preservation (ARP) as well as clinical, radiographic and patient-reported outcomes upon implant placement and crown fabrication at the same site.

Both bone graft materials (FDBA and CEBX) are FDA approved and are widely available in the US market and are routinely used in everyday practices and within the university.

* FDBA is produced by Community Blood Center (Community Tissue Services, Ohio, USA) (FEI: 3008808182).
* CEBX is produced by Geistlich Pharma AG (Wolhusen, Switzerland) [501(k) #: K122894].

Both materials will be stored and utilized based on manufacturers' recommendations and as per of Standard of Care protocols within the university.

Participants and investigators will be unaware of the envelope content and each participant will be asked to randomly pick an envelope and immediately both the participant as well as the investigator will be informed about the envelope content and, therefore, the group allocation. Eventually, participants and investigators will be aware of the group allocation, except for the investigator who will conduct all the study measurements who will remain blinded.

Upon healing, both groups will receive similar treatment as far as implant placement and crown restoration is concerned.

Interventions and procedures

The study-related interventions and procedures will more specifically include:

1. Evaluation of horizontal and vertical ridge dimensional changes as well as contour changes upon standard of care procedures (alveolar ridge preservation) through cone beam computed tomography and intraoral scanning, respectively, after 16 weeks of healing.
2. Determination of the feasibility of prosthetically driven implant placement upon standard of care evaluation of the post-healing cone beam computed tomography, at 16 weeks after ARP.
3. Histological evaluation of the healed grafted area upon grafting with frequently used bone graft materials at 16 weeks of healing.
4. Assessment of peri-implant clinical and radiographic parameters as well as crown esthetics and patient satisfaction upon 12 months from the dental implant placement.

ELIGIBILITY:
Inclusion Criteria:

* patients able to provide informed consent
* patients of 18 years of age or older at time of consent and enrollment
* patients in need of at least one anterior tooth extraction and seeking dental implant replacement
* bone on the buccal of the central/lateral incisors or canines planned for extraction that is either intact or has a dehiscence </=5mm as determined radiographically through cone beam computed tomography (CBCT)

Exclusion Criteria:

* current smokers or tobacco-product users (self-reported)
* uncontrolled diabetes (HbA1c≥7 in the last 3 months)
* pregnant and/or lactating females (self-reported)
* patients on immunosuppressants, steroids, bisphosphonates or other medications that have been related to Medication-Related Osteonecrosis of the Jaw (MRONJ) as described by the American Association of Oral Maxillofacial Surgeons (AAOMS) 2014 update
* patients with history of radiation of the head and neck
* patients with allergy to collagen, bacitracin and/or polymyxin B
* patients with religious or cultural beliefs that prohibit the use of either allograft or bovine graft material
* patients with physical and/or mental/cognitive disabilities (self-reported) or decisionally-impaired, not able to consent for themselves
* patients with untreated periodontitis
* patients with central/lateral incisors or canines requiring extraction and are adjacent to an edentulous area
* patients with central/lateral incisors or canines with buccal bone dehiscence >5mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in radiographic horizontal and vertical ridge dimensions | baseline to 16 weeks after surgery
  Linear radiographic horizontal (HRD) and vertical (VRD) ridge dimensional changes will be measured and compared between groups after 16 weeks of healing.

SECONDARY OUTCOMES:
Mean change in alveolar ridge contour | baseline to 4 weeks after surgery
  Alveolar ridge contour changes as they appear on intraoral optical scans will be measured and compared between groups.
Mean change in alveolar ridge contour | baseline to 2 months after implant placement, approximately 24 weeks
  Alveolar ridge contour changes as they appear on intraoral optical scans will be measured and compared between groups.
Mean change in alveolar ridge contour | baseline to 12 months after implant placement, approximately 70 weeks
  Alveolar ridge contour changes as they appear on intraoral optical scans will be measured and compared between groups.
Number of implants/participants with an implant placed on a prosthetically driven position | 16 weeks
  Feasibility of prosthetically driven implant placement will be assessed with an implant planning software on the cone beam computed tomography obtained at 16 weeks after the ARP, and compared between groups
Mean percentage of residual bone graft particles | 16 weeks
  Histologic evaluation of grafted sites from both groups will be performed at the time of implant osteotomy preparation, 16 weeks upon the ARP surgery.
  Parameters such as residual bone graft particles, new bone formation and connective tissue will be assessed and compared between groups.
Mean percentage of new bone formation | 16 weeks
  Histologic evaluation of grafted sites from both groups will be performed at the time of implant osteotomy preparation, 16 weeks upon the ARP surgery.
  Parameters such as residual bone graft particles, new bone formation and connective tissue will be assessed and compared between groups.
Mean percentage of connective tissue | 16 weeks
  Histologic evaluation of grafted sites from both groups will be performed at the time of implant osteotomy preparation, 16 weeks upon the ARP surgery.
  Parameters such as residual bone graft particles, new bone formation and connective tissue will be assessed and compared between groups.
Mean probing depth | 2 months after implant placement (approximately 24 weeks) and 12 months after implant placement (approximately 70 weeks)
  Probing depths will be recoded at 6 sites on each implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual) with a periodontal probe to the nearest mm. Mean probing depths will be compared between groups at 2 and 12 months after the implant placement.
Mean percentage of implant surfaces with bleeding | 2 months after implant placement (approximately 24 weeks) and 12 months after implant placement (approximately 70 weeks)
  Presence or absence of bleeding upon probing with a periodontal probe will be recoded at 6 sites on each implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). The mean percentage of bleeding will be compared between groups at 2 and 12 months after the implant placement.
Mean percentage of implant surfaces with plaque | 2 months after implant placement (approximately 24 weeks) and 12 months after implant placement (approximately 70 weeks)
  Presence or absence of plaque that can be collected with a periodontal probe will be recoded at 6 sites on each implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). The mean percentage of plaque will be compared between groups at 2 and 12 months after the implant placement.
Mean width of keratinized mucosa | 2 months after implant placement (approximately 24 weeks) and 12 months after implant placement (approximately 70 weeks)
  The width of the keratinized mucosa will be measured to the nearest mm with a periodontal probe on the mid-facial and mid-lingual aspect of each implant. The mean width of keratinized mucosa will be compared between groups at 2 and 12 months after the implant placement.
Mean migration of peri-implant mucosal margin | 2 months after implant placement (approximately 24 weeks) and 12 months after implant placement (approximately 70 weeks)
  The migration of the peri-implant mucosal margin will be measured to the nearest mm with a periodontal probe on the mid-facial and mid-lingual/palatal aspect of each implant. The mean migration of peri-implant mucosal level will be compared between groups at 2 and 12 months after the implant placement.
Mean change peri-implant marginal bone level changes | 16 weeks to 2 months after implant placement (approximately 8 weeks) and 16 weeks to 12 months after implant placement (approximately 54 weeks)
  Peri-implant marginal bone level changes from implant placement to 2 and 12 months after the implant placement will be evaluated and compared through standardized bitewing radiographs.
Mean implant-crown esthetic score | 12 months after implant placement, approximately 70 weeks
  Implant crown esthetics will be evaluated through the Pink Esthetic Score (PES) at 12 months after the implant placement. The PES ranges from 0-12 with higher scores indicating better outcome.
Mean patient satisfaction score | 12 months after implant placement, approximately 70 weeks
  Patient satisfaction will be evaluated and compared with a two-item survey, including the following questions to be answered using the 0-10 Visual Analogue Scale (VAS):
  * "Are you satisfied with the final outcome?"
  * "Would you undergo the same procedure in the future?" Scores range from 0-20 with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Elli Anna Kotsailidi, DDS, MS, Principal Investigator — Eastman Institute for Oral Health, University of Rochester
Locations (1):
- Eastman Institute for Oral Health, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No